CLINICAL TRIAL: NCT04173325
Title: Phase I Feasibility and Safety Study of Nivolumab in Combination With Irinotecan in Relapsed or Refractory Small Cell Lung Cancer (SCLC) Followed by Maintenance Nivolumab
Brief Title: Feasibility and Safety Study of Nivolumab With Irinotecan for Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by the IRB 5/26/22 due to non-compliance
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Nagla Abdel Karim, Professor, Hematology/Oncology, Director of Thoracic Oncology and Phase I Program, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCC-20-009
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Lung cancer; Relapsed lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Nivolumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Irinotecan (Experimental): Drug: Nivolumab 360mg IV Day 1 of each 21 day cycle until disease progression or unacceptable toxicity + Drug: Irinotecan 500mg IV Day of each 21 day cycle for 2 cycles Followed by maintenance nivolumab (without irinotecan)
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO]; Drug: Irinotecan Injection [Camptosar]

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML Intravenous Solution [OPDIVO] — PD-1 inhibitor approved by the US FDA for treatment of patients with lung cancer.
Drug: Irinotecan Injection [Camptosar] — Chemotherapy drug currently FDA approved for treatment of multiple tumors, including small cell lung cancer.

SUMMARY:
This study will determine the frequency of adverse events (side effects) in patients with relapsed or refractory small cell lung cancer (SCLC) when given nivolumab and irinotecan together followed by nivolumab maintenance. This study will test the safety of the study treatments when given together and see what effect (good or bad) it has on participants and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SCLC with known UGT1A genotype.
* Patients who have received at least 1 prior platinum-based chemotherapy.
* Life expectancy of 3 months or more.
* Measurable disease.

Exclusion Criteria:

* Patients with UGT1A polymorphism.
* Currently receiving chemotherapy.
* Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the frequency and severity of adverse events in patients with small cell lung cancer after receiving nivolumab plus irinotecan followed by nivolumab maintenance. | through study completion, an average of 1 year
  CTCAE v.4.0. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Overall response rate | through study completion, an average of 1 year
  Tumor response evaluation with RECIST
Progression-free survival (PFS) | through study completion, an average of 1 year
  PFS as measured from start of therapy till disease progression.
Overall survival (OS) | through study completion, an average of 1 year.
  OS as measured from start of therapy till date of death or last follow up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Nagla A Karim, MD, PhD, Principal Investigator — Augusta University Georgia Cancer Center
Locations (1):
- Georgia Cancer Center at AU Medical Center, Augusta, Georgia, United States